CLINICAL TRIAL: NCT02329483
Title: Early Follicular Phase Androstenedione Monitoring During Low-dose Step-up Induction of Ovulation in High Responders
Brief Title: Monitoring the Early Follicular Phase With Androstenedione in Low-dose Step-up Ovulation Induction in High Responders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Eser Sefik Ozyurek, Operator Doctor, Bagcilar Training and Research Hospital
Other Study IDs: BagcilarTRH
Record Dates: First submitted 2014-12-29; First posted 2014-12-31 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Infertility; Ovarian Hyperstimulation Syndrome
Keywords: Infertility; Ovulation induction; Low-dose step-up protocol; Ovarian high responder; Androgens; Androstenedione; Testosterone; rhFSH
MeSH Terms: conditions — Infertility; Ovarian Hyperstimulation Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- High responder infertile patients: Ovarian high responder patients who are being planned for low-dose step-up protocol ovulation induction and intrauterine insemination.

SUMMARY:
This study aims to predefine the threshold FSH doses during the early follicular phases in low- dose step-up ovulation induction cycles used to treat anticipated high responders by monitoring total testosterone and androstenedione blood levels. The blood levels of total testosterone and androstenedione levels will be measured in patients at the starting day and at every control day when vaginal sonographic folliculometries and blood estradiol measurements are made. Hence, we are aiming to define an early monitoring parameter by which we will be able to define a follicular response to treatment before estradiol rise or apparently selected follicular growth.

DETAILED DESCRIPTION:
50 patients with anticipated high ovarian response, who are being planned to be conventionally treated with low-dose step-up ovulation induction and intrauterine insemination will be analysed in this study. At every control day including the start day, blood samples taken for blood estradiol (and if required progesterone) measurements will be used to measure blood androstenedione and total testosterone levels, as well. Hence, we will have defined an early parameter for defining follicular response in the first 5-7 days of low-dose step-up ovulation induction. Low-dose step-up ovulation induction will be started at 50-75Units/day of rhFSH and the dose will be increased at not earlier than the 7th day at an increment of +37,5Units/day unless a response is observed ( which is at least a 10mm follicle, selected for growth). If more than 3 dominant follicles are selected, the cycle will be cancelled. Otherwise, when at least one follicle >16mm is obtained, a 150Microgram sc. injection will be administered for ovulation trigger and intrauterine insemination made at the 34th-36th hours.

ELIGIBILITY:
Inclusion Criteria:

* Primary/Secondary infertile women; aged 20-35 years of age
* High ovarian response to ovulation induction anticipated.(Antral follicle count on the 3rd day of cycle>10)
* Mild male factor or normal sperm parameters
* Normal anatomic findings with the HSG
* Eugonadotropic
* Normal blood prolactin and TSH levels

Exclusion Criteria:

* Amenorrheic women
* Women with Diabetes Mellitus
* Body Mass Index: <22 or >30
* Age<20 or >35 years old
* Hormonal abnormalities: regarding prolactin, TSH
* Hypo- or Hypergonadotropic women
* Additional medical or surgical disease
* Ovarian cysts
* Previous ovarian surgery

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Primary/Secondary Infertile patients (couples); ovarian high response to ovulation induction anticipated; with mild male factor or without any male factor. Hysterosalpingography reveals patent uterine tubes and normal uterine cavity.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-05 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Blood androstenedione and testosterone levels. | within 10-20 days
  Patterns of blood androstenedione and testosterone levels with respect to the regular monitoring parameters and relations to secondary outcomes.

SECONDARY OUTCOMES:
Pregnancy | 20-30 days
  blood hCG level >10mIU/mlt
Cycle cancellation | within 10-20 days
  cancellation of treatment despite 2 rounds of dose step-up
Ovarian hyperstimulation | 10-30 days
  Enlarged ovaries, abdominal ascites, pleural effusion, hemoconcentration, abdominal swelling
Need for dose step-up | 7-14 days
  if at the 7th day of a dose, no follicle(s)>10mm are observed then the dose is increased

CONTACTS AND LOCATIONS:
Overall Officials: Eser S Ozyurek, MD, Study Director — Bagcilar Training and Research Hospital; Erdal Kaya, Prof Dr, Study Chair — Bagcilar Training and Research Hospital; Mustafa U Karacaoglu, MD, Study Chair — Bagcilar Training and Research Hospital; Evrim E Kovalak, MD, Study Chair — Bagcilar Training and Research Hospital; Erdinc Ergul, MD, Study Chair — Bagcilar Training and Research Hospital
Locations (1):
- Bagcilar Training and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Ozyurek ES, Yoldemir T, Artar G. Androstenedione response to recombinant human FSH is the most valid predictor of the number of selected follicles in polycystic ovarian syndrome: (a case-control study). J Ovarian Res. 2017 May 12;10(1):34. doi: 10.1186/s13048-017-0330-7. PMID 28494798